CLINICAL TRIAL: NCT04924010
Title: Effect of Perioperative Cognitive Behavioural Therapy on Chronic Persistent Postsurgical Pain Among Breast Cancer Patients With High Pain Catastrophising Characteristics: A Randomised, Double-blind Clinical Trial
Brief Title: Effect of Perioperative CBT on Chronic Persistent Postsurgical Pain Among Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Aneurin Moorthy, Research Fellow in Anaesthesia and Perioperative Medicine, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBTMMUH
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Chronic Pain; Chronic Postsurgical Pain; Quality of Life
Keywords: Breast Surgery; Chronic PostSurgical Pain (CPSP); Mastectomy; Wide Local Excision; Cognitive Behavioural Therapy (CBT); Psychological factors; Perioperative; Pain catastrophizing; Anxiety
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Pain, Postoperative; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Educational Status; Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to which intervention they will receive. The outcome assessors for this study will be unaware as to which group the participant will be randomised to and therefore they will be blinded to which intervention the participant had received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (CBT) (Active Comparator): Cognitive behavioural therapy (CBT) is a talking therapy that can help patients manage problems by changing the way they think and behave. It's most commonly used to treat anxiety, depression and chronic pain conditions.
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Education and Mindfulness (Placebo Comparator): Education and mindfulness therapy refers to lessons on techniques to calm the mind and body - can reduce the negative effects of stress
  Interventions: Behavioral: Education and Mindfulness

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — The CBT intervention will be delivered by a Senior Psychologist with seventeen years of hospital psychology experience, six in the treatment of chronic pain patients. Sessions are delivered in one hour, individual therapy appointments to patients, and there is an emphasis on relaxation training, cognitive restructuring, exercise and pacing, behavioral activation, improving sleep, and anger management. Standardized worksheets and homework assignments are an important part of CBT-CP and these will be given (post or email) to patients who will be asked to read and complete in terms of complementing the consultations. This intervention has been developed with reference to two sources: A successful national implementation of CBT for chronic pain (CBT-CP) using video teleconferencing format [Connolly KS et al] AND an evidence-based CBT manual specifically designed to treat chronic pain [Murphy JL et al].
  Arms: Cognitive Behavioural Therapy (CBT)
Behavioral: Education and Mindfulness — To control for differences in attention between the two interventions, patients in the mindfulness group will also have two meetings before the surgery and two meetings afterward. As the same person will be providing the CBT-CP and educational interventions, this confounding factor will be controlled for. The control intervention consists of discussing pain education, as derived from the self-management section of the chronic pain Ireland website (https://www.chronicpain.ie/our-services/self-management) and the persistent pain section of the pain toolkit website (https://www.paintoolkit.org/persistent-pain). Four mindfulness-based stress reduction exercises will be completed including an introductory session on mindful breathing, a guided meditation, progressive muscle relaxation, and a body scan. These sessions will last about half an hour.
  Arms: Education and Mindfulness

SUMMARY:
Chronic persistent post-surgical pain (CPSP) is defined as pain at or near the site of surgery persisting for 3 months or more after the date of surgery. The incidence CPSP in Europe is up to 50% at 3 months and 12% at 12 months, but the incidence varies depending on surgical procedure [Fletcher D et al]. In Breast surgery, one of the most commonly performed surgical procedures for cancer [Kehlet H et al], CPSP has been observed in 20-30% of patients at 6 months after surgery, making this group among the highest risk of developing CPSP [Spivey TL et al & Weiser TG et al]. Clinical developments that could mitigate the development of CPSP after breast cancer surgery would potentially yield multiple benefits in terms of reducing future healthcare utilization, associated costs [Spivey Tl et al], and improving their physical and mental health.

Several predictive factors for CPSP have been identified, the most important being chronic pre-operative pain, high intensity of acute postoperative pain, and several psychological factors [Vranceanu A-M et al]. Of these psychological factors, pain catastrophizing has emerged as one of the strongest predictors of pain severity and disability among individuals with a range of pain presentations and CPSP [Leung L & Wade Jb & Wildeman TH]. Catastrophizing is described as a maladaptive psychological coping strategy involving an exaggerated reaction to anticipated or actual pain. It can involve mental rumination, magnification of the perceived danger or threat associated with pain, and feelings of helplessness in relation to what can be done [Leung L et al]. A recent systematic review on psychological interventions undergoing major elective abdominal surgery concluded catastrophization can have a direct influence on the neuropathophysiological mechanisms underlying pain experiences and can improve pain and psychological outcomes, after surgery [Villa G et al].

In recent years, there has been a growing number of studies investigating the potential impact of perioperative psychological interventions in a variety of patient groups. A recent systematic review and meta-analysis of observational studies concluded that psychological predictors may have a significant association with chronic postsurgical pain, including catastrophization, although this conclusion is limited by the heterogeneity of study designs and methods used [Giusti et al]. To our knowledge, no randomized controlled trial has been done to date, investigating the influence of perioperative psychological interventions on CPSP in patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
This will be a single-center, prospective, double-blinded, randomized controlled trial. The study will randomize breast cancer surgery patients into two groups: one that receives perioperative cognitive-behavioral therapy (CBT) in addition to usual care and the other receives an educational program. The estimated duration for the main investigational plan (e.g. from the start of screening of the first participant to the last participant processed and finishing the study) is one year.

Aims and objectives:

The primary objective is to examine whether a perioperative CBT-based psychological intervention is effective at reducing pain intensity at three-month follow-up, in high catastrophizing patients undergoing breast cancer surgery, compared to an education program.

Secondary objectives of the study include examining whether perioperative CBT has a demonstrable impact on patients, compared to a time-matched education program, with regard to additional self-reported secondary outcomes, including quality-of-recovery, pain catastrophizing, pain interference, depression, and anxiety.

Participants and recruitment:

Adult patients who are undergoing breast surgery (defined as wide excision with magseed surgery or full mastectomy patients with or without axillary clearance) who are proficient in the English language will be eligible for inclusion. Patients will be enrolled at the outpatient clinic of the Department of Anaesthesiology and the Breast Health Department at the Mater Misericordiae University Hospital. All patients entering the screening phase of the study will be registered on a Study Patient Registration Log and a unique registration number will be assigned. Clinical data will be assessed to evaluate a subject's eligibility.

Patients eligible for participation will be evaluated approximately two weeks before surgery and asked for informed consent, and then asked to complete the Pain Catastrophizing Scale (PCS) [Sullivan M et al] by a member of the research team. Patients with high pain catastrophizing, defined as a score of ≥24 on the PCS, will be eligible for randomization to perioperative treatment with CBT or the education and mindfulness program. This cut-off is based on a previous study that showed a pre-treatment score of 24 or higher on the PCS best-predicted follow-up chronic pain ratings and work status after multidisciplinary treatment[Scott W et al] and has since been selected as an appropriate score cut-off in a perioperative CBT intervention in lumbar surgery patients [Scarone P et al]. More recently, this cut-off was also suggested to obtain the highest sensitivity and specificity to predict unfavorable outcomes after spinal surgery [Tuna T et al].

Randomization:

Patients will be randomized after they are included in the study, having consented and completed the PCS (and scoring scored ≥24), and two preoperative appointments will be scheduled with the patients in the intervention and control groups. Patients will be randomized to either 'CBT' or 'Education' group by using an online computer-generated block randomization. The patient study number and group allocation will be typed onto separate pages and concealed in sequentially numbered sealed envelopes. Block randomization will occur as follows; 12 subjects per block to ensure even numbers of participants in each arm of the study and the number of blocks that will be used is 4. Randomization will be performed by an independent third party. The randomization key/seed will also be held by an independent third party and investigators will not have access to this key/seed until the study has been completed.

The envelope will be opened by the treating psychologist to reveal the group allocation. Patients and members of the research team involved in data collection and analyzing the data will be masked to group allocation. The treating psychologist will not be blinded. Group allocations will be revealed immediately if there was a clinical concern.

All patients in both interventional arms:

All patients, irrespective of group allocation, will be routinely prescribed medications for pain control and will be referred for physical therapy on an out-patient basis, or other services, depending on clinical indications and personal needs.

Sample size, power considerations, and statistical analysis:

The primary outcome is the difference in the BPI average pain severity score and average pain interference score between the study groups, three months after surgery. A clinically important difference on the BPI is a 2 raw score reduction on the 11-point NRS [Wong K et al & Marcus J et al & Mease PJ etl al]. The standard deviation (SD) of BPI scores after breast surgery is in the order of 2.3 on this scale (Burckhardt CS et al). Taking a BPI score reduction of 2 as being clinically significant, then n=21 patients would be required each arm if Type I error=0.05 and Type II error is 0.2 (power 80%). Taking into account a 10% drop-outs rate, we propose to enroll 24 eligible patients in each group (N=48 total).

Baseline patient characteristics will be stratified by group and presented as mean and standard deviation (SD), median and first and third quartile, and count and percentage, as appropriate. Differences in baseline characteristics between randomized groups will not be statistically tested, whereas differences with the separate control cohort will be tested using the independent-samples t-test for continuous variables, and Pearson's chi-square test for categorical variables. In case of expected cell counts of less than 5, Fisher's Exact test will be used instead.

All patients randomized (i.e. those with a PCS score > 24) will be analyzed in an intention-to-treat analysis. To test for a difference between the CBT and control group in the BPI 'average' pain intensity scale at three months, linear regression will be used. Adjustment for the type of surgery, age, and education will be made and, if necessary, for other prognostic variables significantly associated with the outcome (i.e., acute postoperative pain intensity, the severity of catastrophizing, preoperative depression, preoperative surgical fear, length of current sick leave, pain duration).

Secondary outcome variables will be analyzed similarly to the primary outcome. For these, logistic regression analysis will be used to test for differences in proportions at three months postoperatively. For exploratory purposes, we will compare the outcomes of the patients in the two intervention groups with the outcomes of patients with low pain catastrophizing scores (i.e. those with a PCS score < 24) undergoing care as usual. Linear mixed-effects regression for the three groups will be performed with primary and secondary outcomes at the three postoperative assessment periods and controlling for preoperative values. This analysis will indicate whether high catastrophizing patients follow a similar trajectory of pain and functioning after breast surgery compared to non-catastrophizing patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* 18-75 years of age
* Undergoing breast cancer surgery (wide local excision with magseed or full mastectomy)
* Pain Catastrophizing Scale score of 24 of higher

Exclusion Criteria:

* Pain Catastrophizing Scale score below 24
* Surgery for benign breast disease
* Patient non-consent
* Plans to undergo major surgery within six months after current breast surgery
* Comorbid severe psychiatric conditions such as schizophrenia or personality disorder
* Known or suspected non-compliance
* Known or suspected drug or alcohol abuse problems within past 3 months
* Inability to follow the study procedures e.g. dementia or non-fluency of English
* The presence of any serious medical comorbidity such as sepsis or cancer that might cause disability or worsen the patient's general health condition
* Pregnancy
* An opioid intrathecal pump
* Prisoner within the criminal justice system
* Cognitive behavioural therapy in the past 12 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Short-form: average pain severity | 3 months post-operative
  BPI Short-form is a 9 item questionnaire used to evaluate the severity of a patient's cancer or non cancer pain [Tan G et al]. Brief Pain Inventory short-form scale is measured between 0 - 10, where '0' indicates no pain and '10' indicates severe pain. A decrease in the Brief Pain Inventory score of 2 or more from the baseline score is considered significant and indicates an improvement in severity of the patient's cancer and non-cancer pain.

SECONDARY OUTCOMES:
Quality of Recovery-15 (QoR-15) Score | 24 hours post-operative
  QoR-15 is a 15-item questionnaire which is used as a tool to assess overall patient recovery and pain after surgery. Participant will be asked to complete this questionnaire within24-48 hours after their surgery. It is scored between 0 and 150, where the greater the number indicates excellent post-operative recovery. [Chazapis M et al].
Pain Catastrophizing Scale (PCS) Score | 3 months post-operative
  PCS is a 13-item questionnaire designed to measure levels of pain-catastrophizing. The scale comprises 13 items which yield an overall catastrophizing score, which is a composite of magnification, rumination, and helplessness subscales [Sullivan M et al]. A Pain Catastrophizing score of greater than 24 is significant for increased risk of developing chronic pain.
Hospital Anxiety and Depression Scale (HADS) Score | 3 months post-operative
  HADS is a 14 item self reported questionnaire that was developed and found to be a reliable method for detecting states of depression and anxiety in the setting of a hospital medical outpatient clinic [Zigmond AS et al]. The score scale ranges between 0-21. A score between 0-7 is normal, a score between 8-10 is considered borderline abnormal and a score between 11-21 is abnormal and indicates a high likelihood that the patient is suffering from anxiety and or depression.
Brief Pain Inventory (BPI) Short-form: average interference score | 3 months post-operative
  BPI Short-form is a 9 item questionnaire used to evaluate the interference the pain has on his/her daily functioning [Tan G et al]. BPI is measured between 0 - 10, where '0' indicates no interference and '10' indicates severe interference with quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Donal Buggy, MB Bch BAO, Principal Investigator — Department of Anaesthesiology & Perioperative Medicine, Mater Misericordiae University Hospital,
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data sharing will be supported with qualified external researchers and supporting clinical documents from eligible studies. All data provided will be coded and anonymised to respect the privacy of patients who have participated in the trial
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: Publications, reports or query requests from future investigators.

REFERENCES:
- [Background] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Spivey TL, Gutowski ED, Zinboonyahgoon N, King TA, Dominici L, Edwards RR, Golshan M, Schreiber KL. Chronic Pain After Breast Surgery: A Prospective, Observational Study. Ann Surg Oncol. 2018 Oct;25(10):2917-2924. doi: 10.1245/s10434-018-6644-x. Epub 2018 Jul 16. PMID 30014456
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Vranceanu AM, Bachoura A, Weening A, Vrahas M, Smith RM, Ring D. Psychological factors predict disability and pain intensity after skeletal trauma. J Bone Joint Surg Am. 2014 Feb 5;96(3):e20. doi: 10.2106/JBJS.L.00479. PMID 24500592
- [Background] Leung L. Pain catastrophizing: an updated review. Indian J Psychol Med. 2012 Jul;34(3):204-17. doi: 10.4103/0253-7176.106012. PMID 23441031
- [Background] Wade JB, Riddle DL, Thacker LR. Is pain catastrophizing a stable trait or dynamic state in patients scheduled for knee arthroplasty? Clin J Pain. 2012 Feb;28(2):122-8. doi: 10.1097/AJP.0b013e318226c3e2. PMID 22001663
- [Background] Wideman TH, Sullivan MJ. Reducing catastrophic thinking associated with pain. Pain Manag. 2011 May;1(3):249-56. doi: 10.2217/pmt.11.14. PMID 24646391
- [Background] Villa G, Lanini I, Amass T, Bocciero V, Scire Calabrisotto C, Chelazzi C, Romagnoli S, De Gaudio AR, Lauro Grotto R. Effects of psychological interventions on anxiety and pain in patients undergoing major elective abdominal surgery: a systematic review. Perioper Med (Lond). 2020 Dec 8;9(1):38. doi: 10.1186/s13741-020-00169-x. PMID 33292558
- [Background] Giusti EM, Lacerenza M, Manzoni GM, Castelnuovo G. Psychological and psychosocial predictors of chronic postsurgical pain: a systematic review and meta-analysis. Pain. 2021 Jan;162(1):10-30. doi: 10.1097/j.pain.0000000000001999. PMID 32694386
- [Background] Scott W, Wideman TH, Sullivan MJ. Clinically meaningful scores on pain catastrophizing before and after multidisciplinary rehabilitation: a prospective study of individuals with subacute pain after whiplash injury. Clin J Pain. 2014 Mar;30(3):183-90. doi: 10.1097/AJP.0b013e31828eee6c. PMID 23552561
- [Background] Scarone P, Smeets AYJM, van Kuijk SMJ, van Santbrink H, Peters M, Koetsier E. A randomized controlled TRIal of cognitive BEhavioral therapy for high Catastrophizing in patients undergoing lumbar fusion surgery: the TRIBECA study. BMC Musculoskelet Disord. 2020 Dec 4;21(1):810. doi: 10.1186/s12891-020-03826-w. PMID 33276768
- [Background] Tuna T, Boz S, Van Obbergh L, Lubansu A, Engelman E. Comparison of the Pain Sensitivity Questionnaire and the Pain Catastrophizing Scale in Predicting Postoperative Pain and Pain Chronicization After Spine Surgery. Clin Spine Surg. 2018 Nov;31(9):E432-E440. doi: 10.1097/BSD.0000000000000694. PMID 30036209
- [Background] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Wong K, Zeng L, Zhang L, Bedard G, Wong E, Tsao M, Barnes E, Danjoux C, Sahgal A, Holden L, Lauzon N, Chow E. Minimal clinically important differences in the brief pain inventory in patients with bone metastases. Support Care Cancer. 2013 Jul;21(7):1893-9. doi: 10.1007/s00520-013-1731-9. Epub 2013 Feb 15. PMID 23411998
- [Background] Marcus J, Lasch K, Wan Y, Yang M, Hsu C, Merante D. An Assessment of Clinically Important Differences on the Worst Pain Severity Item of the Modified Brief Pain Inventory in Patients with Diabetic Peripheral Neuropathic Pain. Pain Res Manag. 2018 Jul 22;2018:2140420. doi: 10.1155/2018/2140420. eCollection 2018. PMID 30140328
- [Background] Mease PJ, Spaeth M, Clauw DJ, Arnold LM, Bradley LA, Russell IJ, Kajdasz DK, Walker DJ, Chappell AS. Estimation of minimum clinically important difference for pain in fibromyalgia. Arthritis Care Res (Hoboken). 2011 Jun;63(6):821-6. doi: 10.1002/acr.20449. PMID 21312349
- [Background] Burckhardt CS, Jones KD. Effects of chronic widespread pain on the health status and quality of life of women after breast cancer surgery. Health Qual Life Outcomes. 2005 Apr 28;3:30. doi: 10.1186/1477-7525-3-30. PMID 15860132
- [Derived] Moorthy A, Lowry D, Edgely C, Blajeva M, Casey MB, Buggy DJ. Perioperative cognitive behavioural therapy compared with pain education and mindfulness for chronic postsurgical pain in breast cancer patients with high pain catastrophising characteristics: a randomised, controlled, parallel group clinical trial. BJA Open. 2025 Oct 30;16:100499. doi: 10.1016/j.bjao.2025.100499. eCollection 2025 Dec. PMID 41234748
- [Derived] Moorthy A, Lowry D, Edgley C, Casey MB, Buggy D. Effect of perioperative cognitive behavioural therapy on chronic post-surgical pain among breast cancer patients with high pain catastrophising characteristics: protocol for a double-blinded randomised controlled trial. Trials. 2022 Jan 21;23(1):66. doi: 10.1186/s13063-022-06019-z. PMID 35062997
- See also: Nationwide implementation and outcomes of cognitive behavioral therapy for chronic pain over clinical video teleconferencing. J Technol Behav Sci — https://doi.org/10.1007/s41347-017-0024-4
- See also: Cognitive behavioral therapy for chronic pain among veterans: therapist manual. Washington, DC: Department of Veterans Affairs — https://www.va.gov/painmanagement/docs/cbt-cp_therapist_manual.pdf
- See also: Pain education, self-management section of the chronic pain Ireland — https://www.chronicpain.ie/our-services/self-management